CLINICAL TRIAL: NCT05260190
Title: Hand Grip Strength and Manual Dexterity Modifications After Application of Transcranial Static Magnetic Field Stimulation (tSMS) Over the Primary Motor Cortex (M1) in Healthy Subjects
Brief Title: Manual Dexterity Modifications After Application of tSMS Over the Primary Motor Cortex (M1)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Principal Investigator, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: URJCtSMS100222
Record Dates: First submitted 2022-02-10; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Stroke; Neurologic Disorder; Manual Dexterity
MeSH Terms: conditions — Stroke; Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Several devices (helmets) were available for the active and sham intervention. An investigator outside the study intervention labeled the active and sham helmets with an alphabetic code (A or B). The investigator applying the stimulation did not know which type of intervention was applying (A or B). Neither the investigator performing the intervention, nor the participant knew which intervention corresponded to each group. The data were analyzed by another researcher who was not involved in the assignment and intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tSMS (Experimental): Real tSMS stimulation.
  Interventions: Device: tSMS
- Sham tSMS (Sham Comparator): Sham tSMS stimulation.
  Interventions: Device: Sham tSMS

INTERVENTIONS:
Device: tSMS — 30-minute tSMS application in a comfortable seated position. The material used in the stimulation was a MAGxx1.1 helmet (Neurek Spain Toledo), with a Neodymium (NdFeB) magnet of 60mm diameter and 30mm height with Nickel (Ni-Cu-Ni) coating MAG60r+ (Neurek Spain, Toledo), placed over the primary motor cortex (M1) of the left cerebral hemisphere.
  Arms: tSMS
Device: Sham tSMS — 30-minute sham tSMS application in a comfortable seated position. The device used in sham stimulation had the same weight and shape as the real stimulation helmet.
  Arms: Sham tSMS

SUMMARY:
Transcranial static magnetic field stimulation (tSMS) is a novel brain stimulation technique that has been shown to be safe and effective in modifying biological parameters when applied to the cerebral cortex. Its application decreases cortical excitability, regardless of the polarity of the magnetic field, reducing the amplitude of motor evoked potentials (MEP). tSMS is presented as a potentially useful tool in the management of the interhemispheric inhibition, a condition present in neurological pathologies such as stroke or multiple sclerosis. Despite having demonstrated neurophysiological effects in previous studies, the effects of tSMS application on force production and manual dexterity, have not yet been clearly established.

The present study aims to evaluate changes in force production, manual dexterity, and fatigue after unilateral application of a tSMS session on the primary motor cortex (M1). It is hypothesized that the application of tSMS will momentarily decrease the parameters of strength and manual dexterity in the upper limb contralateral to the stimulated cortex, without changes in the strength and dexterity of the unstimulated hemibody. These parameters may show an increase in the unstimulated hemibody. If the hypothesis is confirmed, it could be considered a valid treatment for health conditions presenting interhemispheric inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years.
* Absence of cognitive impairment.
* Adequate understanding of verbal and written information, sufficient to complete the tests.

Exclusion Criteria:

* Presence of metallic implants (e.g., neurostimulator, pacemaker, cochlear implant, or metallic elements in the head or around the eyes).
* Diagnosis of epilepsy or being under treatment with antiepileptic drugs.
* Diagnosis of unstable cardiovascular disease.
* Diagnosis of any disease or condition that may interfere with this study.
* Use of drugs that may influence with neuromuscular function (muscle relaxants or some analgesics...).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Finger Tapping Test (FTT) | 5 minutes
  was performed for assessment of manual motor skills. This test has been used for many years in the neuropsychological assessment of brain damage, being an indicator of cortical activity, as well as being used in NIBS studies as a measure of manual dexterity.
Nine-Hole Peg Test (9HPT) | 5 minutes
  Was used to assess finger dexterity; this tool has been used in the assessment of motor activity in a multitude of pathologies, with adequate to excellent inter-rater reliability and excellent inter-rater reliability in healthy adults.

SECONDARY OUTCOMES:
Hand grip strength | 5 minutes
  Upper extremity force production was assessed by grip testing; a hand-held dynamometer (Jamar Plus+; Sammons Preston, Rolyon, Bolingbrook, IL) was used for this purpose. Greater hand grip strength corresponds with greater activation in M1, premotor area (PMA), and supplementary motor area (SMA) in the dominant hemisphere, and of the SMA in the nondominant hemisphere, and may provide information about the functionality of the human brain.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes